CLINICAL TRIAL: NCT01597206
Title: Outcomes of Interventions for Patients With a Reduced Posterior Dental Arch: A Randomized Controlled Trial
Brief Title: Interventions for Patients With a Shortened Dental Arch
Acronym: SDA-RCT
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of the Western Cape (Other)
Responsible Party: Principal Investigator, Dr Saadika Khan, Dr, University of the Western Cape
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SDA Clinical Trial; SDA South African RCT (Other: UWC- SA)
Record Dates: First submitted 2012-05-09; First posted 2012-05-11 (Estimated); Last update posted 2017-02-13 (Actual); Status verified 2016-01

CONDITIONS: Anomaly of Dental Arch
Keywords: randomized controlled trial; intervention; posterior reduced dental arch; patient satisfaction; sequential sampling
MeSH Terms: conditions — Patient Satisfaction | interventions — Denture, Partial, Removable

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Removable partial denture Group (Experimental): Patients with a reduced posterior dental arch will be randomized into one of 2 Groups Group A will receive a removable partial denture prosthesis
  Interventions: Device: Removable partial denture (Chrome Cobalt Distal extension)
- Reduced Posterior Dental Arch Group (Active Comparator): Patients with a reduced posterior dental arch and not receiving any Intervention will be compared to the removable partial denture group
  Interventions: Other: A reduced posterior dental arch

INTERVENTIONS:
Device: Removable partial denture (Chrome Cobalt Distal extension) — For Group A: a distal extension removable denture will be constructed for patients with a reduced posterior dental arch
  Other Names: Chrome Cobalt Distal extension denture for Group A patients
  Arms: Removable partial denture Group
Other: A reduced posterior dental arch — For Group B: Patients with a reduced posterior dental arch will not be provided with a removable denture and will be compared to patients in Group A
  Other Names: No intervention for Group B patients
  Arms: Reduced Posterior Dental Arch Group

SUMMARY:
Dental services for large sectors of the population of the Western Cape (WC) Province of South Africa (SA) has been, and continues to be, limited to low-cost treatment options and emergency services, such as extractions at public health clinics. Replacement of missing teeth for the disadvantaged majority of the population is provided almost exclusively at the dental teaching institutions. Loss of teeth in the WC Province is, as elsewhere, the result of disease and the lack of restorative care and then having these replaced by a removable partial denture, if the patient can afford it Null Hypothesis: The daily functional needs and quality of life of partially dentate adult patients with a reduced posterior dental arch and /or a Shortened Dental Arch (SDA) will not be satisfied nor improved by replacing the posterior teeth with a removable prosthesis.

DETAILED DESCRIPTION:
The aim of this research is to determine whether the daily functional needs and the quality of life of partially dentate adult patients with a reduced posterior dental arch will be satisfied and improved without having the posterior teeth replaced with a removable prosthesis, as compared to having the use of such prosthesis.

Objectives: To conduct a randomized controlled trial amongst partially dentate adult patients with a reduced posterior dental arch (3-5 pairs of posterior occluding pairs of teeth) and where these patients will be randomly assigned to one of two groups: one group would be provided with a metal- based removable partial denture (RPDP) to replace the posterior teeth, the other will receive no treatment.

Daily functioning ability and patient satisfaction between the groups (with/without RPDP) would then be compared.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Classic SDA
* Patients with a reduced posterior dental arch (from 3-5 posterior occluding teeth)
* Specific Age limits
* Remaining teeth periodontally sound
* Lost molars in one jaw
* Both canines and one premolar should be present

Exclusion Criteria:

* Exclude patients with Angle Class 2 or 3
* Signs of Temporo-mandibular disorders
* Compliance is a problem (Alcoholism/ drug addiction)
* Risk of over-eruption of teeth
* Patients wanting removable partial dentures

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2014-01; Primary Completion 2016-10 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Patient satisfaction | 3 months
  Two different tools will b used to assess primary outcomes
  1. Oral Impact of Daily Performance (OIDP) tool
  2. Global Visual Analogue Scale (VAS)

SECONDARY OUTCOMES:
Functioning | 3 months
  Failure of intervention or patient unhappy with treatment prescribed
Oral health-related Quality of Life | 3 months
  A Tool will be used to assess primary outcome

OTHER OUTCOMES:
Negative outcomes with intervention | 3 months
  These include: periodontal breakdown (plaque index, loss of attachment), tooth loss, carious lesion formation, change in treatment or any other self-reported complaints

CONTACTS AND LOCATIONS:
Overall Officials: Saadika Khan, PhD, Principal Investigator — Staff Member
Locations (1):
- Saadika Khan, Cape Town, Western Cape, South Africa

IPD SHARING:
Plan to Share IPD: Yes
By publishing the results in a reputable (peer reviewed and accredited) journal